CLINICAL TRIAL: NCT00172809
Title: A Pilot Study in Comparing the Efficacy and Safety of Peginterferon Alfa-2a and Interferon Alfa-2a in Treating Patients With End Stage Renal Disease and Chronic Hepatitis C
Brief Title: Interferon Treatment for Patients With Chronic Hepatitis C and End Stage Renal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 940209
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2007-06

CONDITIONS: Chronic Hepatitis C; End Stage Renal Disease
Keywords: Chronic Hepatitis C; End stage renal disease; Hemodialysis; Interferon; Pegylated interferon
MeSH Terms: conditions — Hepatitis C, Chronic; Kidney Failure, Chronic | interventions — peginterferon alfa-2a; Syringes; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Peginterferon alfa-2a (Pegasys, Hoffmann-LaRoche) 135 ug/week for 24 weeks
  Interventions: Drug: Peginterferon alfa-2a
- 2 (Active Comparator): Interferon alfa-2a (Roferon, Hoffmann-LaRoche) 3 MU tiw for 24 weeks
  Interventions: Drug: Interferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a 135 ug/week for 24 weeks
  Other Names: Pegasus 135 ug/syringe
  Arms: 1
Drug: Interferon alfa-2a — Interferon alfa-2a 3 MU tiw for 24 weeks
  Other Names: Roferon 3 MU/syringe
  Arms: 2

SUMMARY:
The treatment response with conventional interferon alpha alone in patients with end stage renal disease and chronic hepatitis C is about 33-39%. However, the drop-out rate is 17-29.6%. Pegylated interferon alpha, a newly developed form of interferon with superior pharmacokinetic profiles, has not been used to treatment these patients. We expect the better treatment response treated with peginterferon alpha than conventional interferon. In addition, we also observe the safety of the two drugs during the study. The goal of the study is to compare the efficacy and safety of the two different treatment regimens in patients with chronic hepatitis C and end stage renal disease.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is common among patients with end stage renal disease (ESRD), with the reported prevalence ranging from 8 to 20% in dialysis patients in developed world. In Taiwan, the estimated prevalence of HCV infection in patients with ESRD who maintain hemodialysis ranges from 20 to 24.7%. Although most studies have provided mild to moderate disease activity and a high proportion of normal alanine aminotransferase (ALT) levels, the frequency of bridging hepatic fibrosis or cirrhosis ranges from 5 to 32%. Several studies have shown that chronic hepatitis C adversely affects the survival in patients with ESRD. After renal transplantation, recipients with HCV have an increased risk of liver-related mortality and morbidity compared with those without HCV. Therefore, eradication of HCV can improve clinical outcome in dialysis patients as well as in patients awaiting renal transplantation.

Combined interferon and ribavirin is the standard therapy in HCV-infected patients with normal renal function. However, ribavirin, which is cleared by the kidneys, may cause severe hemolytic anemia and be dangerous in dialysis patients. Two recent meta-analyses showed that the sustained virological responses were (SVR) 39% and 33%; the drop-out rate were 17% and 29.6% in HCV-infected dialysis patients treated with interferon-alpha 3 MU thrice weekly of varied duration. The response and the drop-out rate were higher than that reported in HCV-infected patients with normal renal function (SVR of 7-16% by interferon-alpha 3 MU thrice weekly for 24 weeks; drop-out rate of 5-9%) due to a lower interferon clearance rate.

Peginterferon alpha-2a (40KD) is a modified form of interferon alpha-2a consisting of a branched polyethylene glycol (PEG) chain covalently bound to interferon alpha-2a. A better response of peginterferon alpha-2a than interferon alpha-2a has been demonstrated in HCV-infected patients with normal renal function, either combined with ribavirin or not, due to the superior pharmacokinetic profiles. The clearance of peginterferon alpha-2a for ESRD patients was about 30-40% lower than that in healthy subjects. A similarly pharmacokinetic profile of peginterferon alpha-2a is observed with 135 μg weekly in dialysis patients compared with 180μg weekly in patients with normal renal function.

We expect that peginterferon alpha-2a is superior to interferon alpha-2a in achieving an increased SVR and decreased drop-out rate in dialysis patients. The goal of the study is to compare the efficacy and safety of the two different treatment regimens in patients with chronic hepatitis C and end stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65 years old
* Creatinine clearance (Ccr) < 10 ml/min/1.73 m2
* Receiving regular hemodialysis
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive > 6 months
* Detectable serum HCV-RNA (Cobas Amplicor HCV Monitor v2.0, Roche Molecular Systems, Pleasanton, CA) with dynamic range 600~<500,000 IU/ml

Exclusion Criteria:

* Neutropenia (neutrophil count, <1,500/mm3)
* Thrombocytopenia (platelet <90,000/ mm3)
* Co-infection with HBV or HIV
* Chronic alcohol abuse (daily consumption > 20 g/day)
* Decompensated liver disease (Child classification B or C)
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Sustained histological response and sustained virological response 6 months after the completion of the intervention | 1 year

SECONDARY OUTCOMES:
The overall tolerance of the two different regimens and the comparison of the rates of side effects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, M.D., Principal Investigator — Department of Internal Medicine, National Taiwan Univeristy Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Yun-Lin Branch, Douliu, Taiwan

REFERENCES:
- [Background] Fabrizi F, Dulai G, Dixit V, Bunnapradist S, Martin P. Meta-analysis: interferon for the treatment of chronic hepatitis C in dialysis patients. Aliment Pharmacol Ther. 2003 Dec;18(11-12):1071-81. doi: 10.1046/j.1365-2036.2003.01780.x. PMID 14653826
- [Background] Russo MW, Goldsweig CD, Jacobson IM, Brown RS Jr. Interferon monotherapy for dialysis patients with chronic hepatitis C: an analysis of the literature on efficacy and safety. Am J Gastroenterol. 2003 Jul;98(7):1610-5. doi: 10.1111/j.1572-0241.2003.07526.x. PMID 12873587
- [Background] Huraib S, Iqbal A, Tanimu D, Abdullah A. Sustained virological and histological response with pretransplant interferon therapy in renal transplant patients with chronic viral hepatitis C. Am J Nephrol. 2001 Nov-Dec;21(6):435-40. doi: 10.1159/000046646. PMID 11799259
- [Background] Casanovas-Taltavull T, Baliellas C, Benasco C, Serrano TT, Casanova A, Perez JL, Guerrero L, Gonzalez MT, Andres E, Gil-Vernet S, Casais LA. Efficacy of interferon for chronic hepatitis C virus-related hepatitis in kidney transplant candidates on hemodialysis: results after transplantation. Am J Gastroenterol. 2001 Apr;96(4):1170-7. doi: 10.1111/j.1572-0241.2001.03697.x. PMID 11316166
- [Background] Tokumoto T, Tanabe K, Ishikawa N, Simizu T, Oshima T, Noguchi S, Gouya N, Nakazawa H, Hashimoto E, Fuchinoue S, Hayashi N, Toma H. Effect of interferon-alpha treatment in hemodialysis patients and renal transplant recipients with chronic hepatitis C. Transplant Proc. 1999 Nov;31(7):2887-9. doi: 10.1016/s0041-1345(99)00603-x. No abstract available. PMID 10578327
- [Background] Huraib S, Tanimu D, Romeh SA, Quadri K, Al Ghamdi G, Iqbal A, Abdulla A. Interferon-alpha in chronic hepatitis C infection in dialysis patients. Am J Kidney Dis. 1999 Jul;34(1):55-60. doi: 10.1016/s0272-6386(99)70108-3. PMID 10401016
- [Background] Djordjevic V, Kostic S, Stefanovic V. Treatment of chronic hepatitis C with interferon alpha in patients on maintenance hemodialysis. Nephron. 1998;79(2):229-31. doi: 10.1159/000045035. No abstract available. PMID 9647511
- [Background] Simsek H. Interferon-alpha treatment of haemodialysis patients with chronic viral hepatitis and its impact on kidney transplantation. Nephrol Dial Transplant. 1996 May;11(5):912-3. doi: 10.1093/oxfordjournals.ndt.a027441. No abstract available. PMID 8671933
- [Background] Raptopoulou-Gigi M, Spaia S, Garifallos A, Xenou P, Orphanou H, Zarafidou E, Petridou P, Vrettou H, Vagionas G, Galaktidou G, et al. Interferon-alpha 2b treatment of chronic hepatitis C in haemodialysis patients. Nephrol Dial Transplant. 1995 Oct;10(10):1834-7. PMID 8592590
- [Background] Casanovas Taltavull T, Baliellas C, Sese E, Iborra MJ, Benasco C, Andres E, Gonzalez MT, Gil-Vernet S, Casanova A, Casais LA. Interferon may be useful in hemodialysis patients with hepatitis C virus chronic infection who are candidates for kidney transplant. Transplant Proc. 1995 Aug;27(4):2229-30. No abstract available. PMID 7652784
- [Background] Ozyilkan E, Simsek H, Uzunalimoglu B, Telatar H. Interferon treatment of chronic active hepatitis C in patients with end-stage chronic renal failure. Nephron. 1995;71(2):156-9. doi: 10.1159/000188705. PMID 8569947
- [Background] Barril G, Schez Tomero JA, Garcia Buey L, Motellon JL, Bernis C, Traver JA. Response to alpha 2B interferon (IFN) treatment in a haemodialysis patient with chronic hepatitis C. Nephrol Dial Transplant. 1994;9(9):1354-5. No abstract available. PMID 7816309
- [Derived] Prabhu AR, Rao IR, Nagaraju SP, Rajwar E, Venkatesh BT, Nair N S, Pai G, Reddy NP, Suvarna D. Interventions for dialysis patients with hepatitis C virus (HCV) infection. Cochrane Database Syst Rev. 2023 Apr 25;4(4):CD007003. doi: 10.1002/14651858.CD007003.pub3. PMID 37096802